CLINICAL TRIAL: NCT04641611
Title: Effect of Venous Cannulation Technique on the Incidence of Post-operative Atrial Fibrillation in Patients Undergoing Elective Coronary Artery Bypass Grafting. A Pilot Randomized Controlled Trial.
Brief Title: Effect of Venous Cannulation on the Incidence of Atrial Fibrillation in Patients Undergoing Coronary Artery Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Jean-Francois Morin (Other)
Responsible Party: Sponsor-Investigator, Dr. Jean-Francois Morin, Surgical director, Division of Cardiac and Vascular surgery and Cardiology, Jewish General Hospital
Organization: Jewish General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 000
Record Dates: First submitted 2020-11-11; First posted 2020-11-24 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Coronary Artery Bypass; Cardiac surgery; Risk Factors
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient will be blinded with regards to type of venous cannulation performed intra-operatively.
  Measurement of outcome will be performed by an independent cardiologist, who is blinded to treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cavoatrial cannulation (Active Comparator): Cannulation of the atrium with 2-stage venous cannula.
  Interventions: Other: Cavoatrial cannulation
- Bicaval cannulation (Experimental): Cannulating the superior and inferior vena cavae with separate cannulas, inserted through 2 separate incisions in the right artium going into the superior and inferior vena cavae. No slush added. This technique is used in Right heart procedure (Pulmonic and tricuspid valve) and mitral valve procedures.
  This technique is not routinely used in CABG operations.
  Interventions: Other: Bicaval cannulation

INTERVENTIONS:
Other: Bicaval cannulation — Cannulation of SVC and IVC through right atrium in patients undergoing CABG. with snares applied
  Arms: Bicaval cannulation
Other: Cavoatrial cannulation — Cannulating the right atrium and Inferior vena cava with a 2-stage cannula
  Arms: Cavoatrial cannulation

SUMMARY:
Context Atrial fibrillation is the most frequent arrhythmia following coronary artery bypass grafting. POAF is associated with worse outcomes following CABG. In addition, recurrence of AF is associated with longer hospital stay and higher rate of neurological and renal complications compared to a single episode of AF Objective To estimate the proportion of eligible people who are willing to participate, number of participants who drop out of the trial and use the results of this study to inform a larger study.

Study Design:

Pilot randomized controlled trial. Patients will be blinded to the intervention.

Participants:

The study population will include 40 patients. Patients admitted to the Jewish General Hospital for elective coronary artery bypass grafting from May 2021 will be included in the study. Patients will be included if they were in sinus rhythm with a HR ≥50 bpm, undergoing on-pump coronary artery bypass grafting and hemodynamically stable. Patients will be excluded from the study if they meet any of the following criteria: Second or third degree heart block, LVEF <35%, left atrial volume index ≥42 ml/m2, right atrial volume index > 47 ml/m2, any degree of tricuspid regurgitation, any degree of right ventricular dysfunction, emergency or minimally invasive operation, concurrent valve operation, history of atrial fibrillation or previous cardiac surgery

Study Interventions and Measures Patients will be randomly assigned to one of two treatment groups according to the venous cannulation technique used during surgery. Group A will undergo cavoatrial cannulation with a 2-stage venous cannula. Group B will undergo bicaval cannulation with snares. Similar surgical methods will be used in all treatment groups .

The primary endpoint will be defined as any episode of atrial fibrillation in any participant lasting >5 minutes in duration or any episode leading to hemodynamic compromise (SBP<90 mmHg) or causing symptoms (angina or dyspnea). Atrial fibrillation will be diagnosed using telemetry and a 12-lead ECG. Patients will be followed up in 1 month with a 12-lead ECG to determine their rhythm. The secondary endpoints are the development of RV dysfunction, tricuspid regurgitation and any increase in left atrial volume index as detected by post-operative transthoracic echocardiography.

DETAILED DESCRIPTION:
.Introduction

Atrial fibrillation is the most frequent arrhythmia following coronary artery bypass grafting. Its incidence following cardiac surgery is estimated to be between ~10-60%1-5 . The incidence is lower in patients undergoing isolated coronary artery bypass grafting (~25-30%) compared to valve operations 2,6,7. It most commonly occurs in the first four days following cardiac surgery1,5,8. Despite many efforts to predict and prevent postoperative AF, the incidence has not changed over the past decades1-5,9 .

Although in the past it was thought of as a benign self-limiting complication9, atrial fibrillation after cardiac surgery has been shown to be associated with worse outcomes compared to patients who remain in sinus rhythm postoperatively. It leads to increased length of hospital and ICU stay, higher rate of stroke, wound infection, renal failure, myocardial infarction and has a significant effect on early and long-term mortality2-4. In addition, recurrence of AF is associated with longer hospital stay and higher rate of neurological and renal complications compared to a single episode of AF 5.

1.2Mechanisms of POAF

Several studies have investigated the underlying mechanisms involved in development of post-operative atrial fibrillation. However, these mechanisms remain largely unclear. It is believed that atrial fibrillation is caused by reentry of multiple wavelets of excitation in the presence altered atrial refractoriness. This makes ectopic beats originating from foci in the pulmonary veins more likely to trigger an episode of atrial fibrillation 10-12.

In their comprehensive review, Maesen B et al illustrate the various factors that lead to the development of atrial fibrillation. It is triggered by an interaction of acute factors of surgery and pre-existing factors chronic in the patient 1. In other words, factors related to cardiac surgery such as inflammation, oxidative stress and sympathetic activation, together with the presence of an atrial substrate, predispose to the development of POAF 1,12. The most common co-morbid conditions the increase the susceptibility of AF are hypertension, heart failure, mitral valve disease and coronary artery disease12. These co-morbidities also lead to atrial dilation, which is a key factor in the development of an atrial substrate12.

To support this hypothesis, Maesen B et al explain that drugs, which increase sympathetic activity in the heart such as milrinone, dobutamine and dopamine, increase the incidence of POAF. They also demonstrate that perioperative beta-blockers reduced POAF incidence. This is supported a meta-analysis of 33 randomized controlled trials investigating beta-blocker treatment for prevention of POAF. Perioperative beta-blockers led to a reduction in the incidence of postoperative AF13 .

Maesen B et al also argue that inflammation and oxidative stress -caused by surgical trauma and use of cardiopulmonary bypass- contribute to the development of POAF by demonstrating that treatment with ascorbic acid or N-acetyl cysteine, both antioxidants, reduced the incidence of POAF1.

In addition, drugs with anti-inflammatory properties such as corticosteroids and statins have -in many studies- reduced the incidence of POAF1. This is also supported by various studies that found an association between AF and high levels of inflammatory markers such as C-reactive protein and Interleukin-614.

1.3Risk factors for POAF

Several studies have investigated the risk factors that could lead to the development of postoperative AF and attempted to provide a risk stratification model5,15-17. These attempts were unsuccessful in establishing a comprehensive predictive model for POAF.

The most consistent preoperative risk factor for POAF in those studies is older age 5,15-17. Age has been shown to be most strongly associated with development of POAF. The studies frequently mention the following as pre-operative factors: prior history of AF, congestive heart failure, COPD, diabetes mellitus, left ventricular hypertrophy and left atrial enlargement.

In their prospective study of patients undergoing cardiac surgery, Chu et al found that a CHADS-VASc score of more than 2 (Congestive heart failure, Hypertension [blood pressure >140/90 mmHg or treated hypertension on medication], Age >75years, diabetes mellitus, prior Stroke or transient ischemic attack or thromboembolism, vascular disease, Age 65 to 74 years, Sex category [female gender]) was associated with increased incidence of POAF 17.

Perrier et al confirmed these findings in their cohort study of 1481 patients who underwent isolated CABG8. Additionally, they have found that obesity, renal failure, preoperative beta-blockers and preoperative antiplatelet therapy to be independent risk factors for POAF 8. This is in contrast to most studies, which found that preoperative beta-blockers decreased the incidence of POAF.

In a study by Avi et al, pre-operative right ventricular dysfunction as measured by RV myocardial performance index (MPI) -which is a measurement of RV systolic and diastolic function- was demonstrated to be a predictor of POAF in patients undergoing isolated CABG6.

With regards to postoperative factors, a multicenter observational study found that postoperative withdrawal of beta-blockers or ACE inhibitors correlate with increased incidence of POAF 5.

The role of potassium and magnesium supplementation to treat hypokalemia and hypomagnesaemia in order to prevent ventricular arrhythmias after myocardial infarction is well recognized. In addition, low serum magnesium has been shown to be associated with increased incidence of atrial fibrillation in the general population18. However, low serum magnesium hasn't been well established as a predictor of POAF 19,20. The findings of studies on the beneficial effects of prophylactic administration of magnesium to prevent atrial fibrillation post cardiac surgery have been conflicting.13,21-23 A meta-analysis of 35 RCTs by Fairly et al found that magnesium supplementation reduced the risk of atrial fibrillation postoperatively21. However, their analysis was limited by significant heterogeneity between the studies. While another meta-analysis failed to show a prophylactic effect of magnesium or potassium supplementation against PAOF22 . Cook et al performed a meta-analysis of 5 RCTs after excluding the trials with methodological problems; they failed to show a prophylactic effect of magnesium against AF23.

Furthermore, Kalus et al and Matsuura et al investigated the impact of volume overload on the incidence of AF, they found that increased fluid balance on the first or second postoperative days after cardiac surgery was an independent predictor of POAF 24,25. Both studies hypothesized that volume overload will lead to left atrial dilation and thus predispose to AF. However, neither of the studies had recorded measurements of left atrial size.

Few studies have investigated the intraoperative factors of POAF. It is known that concurrent valve surgery increases the risk of POAF5,17. Other risk factors found consistently in the literature include cardiopulmonary bypass and aortic cross clamp times10,15,16,26. A multicenter study found that bicaval cannulation and pulmonary vein venting might be associated with increased risk of POAF 5. In addition, an earlier retrospective study found that snared bicaval cannulation was associated with increased incidence of postoperative atrial arrhythmias in patients receiving high volume crystalloid cardioplegia. However this effect was not observed when low volume cardioplegia was used to compare unsnared bicaval cannulation with cavoatrial cannulation9.

It has been postulated that atrial incision and atrial ischemia during surgery lead to alterations of atrial conduction and refractoriness thereby predisposing to the development of POAF 10. In addition, Tchervenkov et al found an association between persistence of residual atrial electrical activity during cardioplegic arrest and post-operative atrial tachyarrhythmia27. It might be that atrial activity during cardioplegic arrest -which could be due to inadequate atrial protection - resulted in atrial ischemia, which in turn contributes to POAF development 27. It has been demonstrated that return of relatively warm venous blood to the right atrium and ventricle may lead to myocardial warming thereby diminishing the protective effect of cardioplegia. Older animal studies have shown conflicting results regarding the optimal cannulation technique to reduce myocardial rewarming during arrest28,29. Furthermore, no study prospectively investigated the effect of different cannulation techniques on post-operative atrial tachyarrhythmia.

Due to the scarcity of data regarding the intraoperative risk factors of POAF, these factors are not well recognized and preventative strategies are therefore not well established.

2 Objectives To estimate the proportion of eligible people who are willing to participate, the number of participants who drop out of the trial and use the results of this study to inform a larger study.

3. Study design 3.1 Recruitment and sample size Participants will be screened to enter the study in clinic by the principal investigator who is cardiac surgeon. Only the principal investigator's patients who meet inclusion criteria will be considered in the study. Eligibility to enter the study will be determined during the patient's consultation in clinic.

Considering we usually operate on 1 or 2 patients per week who meet inclusion criteria. We believe that 20 patients per group is reasonable to assess feasibility of recruitment and protocol implementation.

3.2 Study population and study procedure

Patients admitted to the Jewish General Hospital for elective coronary artery bypass grafting from January 2021 will be included in the study. Patients will be screened in clinic prior to admission. The study population will include 40 patients that will be randomly assigned to one of two treatment groups according to the venous cannulation technique used during surgery. Group A will undergo cavoatrial cannulation with a 2-stage venous cannula. Group B will undergo bicaval cannulation with snares.

3.3 Intervention Bicaval cannulation will be performed through in the right atrium. Small tapes are passed around the SVC and IVC. Two purse string sutures are placed in the superior and inferior portions of right atrium. Two small incisions are made inside the purse string sutures. The SVC and IVC are cannulated through the superior and inferior incisions respectively. The purse string sutures and small tapes passed through small tubes and snared. The small tapes snare will act as a tourniquet to prevent venous return to the right atrium. Bicaval cannulation is performed in cases of mitral and tricuspid valve operations to provide a bloodless operative field, superior drainage of venous blood and potentially better protection of the heart compared to cavoatrial cannulation. Similar surgical methods will be used in all treatment groups. We will use a standard sternotomy incision to access the heart, the distal ascending aorta be will cannulated. Antegrade Del Nido cardioplegia will be used to arrest the heart under normothermia. The left internal mammary artery will be grafted to the left anterior descending artery. For the other grafts, the left radial artery and saphenous venous grafts will be used where appropriate. The saphenous vein will be harvested endoscopically and the radial artery will be harvested using an open technique. Pre-operative beta-blockers will be continued to the day of surgery and re-started on the first post-operative day if heart rate and blood pressure were permissible.

3.4 Randomization and blinding Patients will be screened in clinic. They will be blinded to their treatment and will be prospectively randomized on hospital admission by simple randomization using a random numbers table. Randomization will be performed by the principal investigator.

3.5 Study measurements Patients' data, including demographics, number of diseased coronary arteries and comorbidities such as presence of hypertension, chronic kidney disease, diabetes mellitus, peripheral vascular disease, previous stroke or myocardial infarction will be collected. Operative data including patients' temperature, cardiopulmonary bypass time, cross-clamp time, aortic and venous cannulation technique, number and location of bypasses will also be collected. Echocardiographic parameters will be collected preoperatively, intra-operatively and post-operatively. These will include left ventricular ejection fraction, right ventricular function, left and right atrial volume indices, RV myocardial performance index (MPI) and the presence of valvular heart disease. Postoperative data will include serum electrolytes, cardiac biomarkers, volume status and beta-blocker use. Postoperative echocardiogram will be done between POD 3-5 and while the heart is in sinus rhythm and with a heart rate <100bpm whenever possible.

3.8 Data reporting Baseline and demographic data will be summarized by standard descriptive summaries e.g. means and standard deviations for continuous variables and percentages for categorical variables. Hypothesis testing will not be performed as this is a feasibility study and the sample size to too small to yield significant conclusions.

4. Confidentiality Informed consent will be taken in clinic by the principal investigator during participant's visit. Participants will be informed that they're able to withdraw from the study at anytime pre-operatively. An additional consent form separate from the regular operation consent form will be used for the study.

Data will be collected in a paper data collection form which will then be transferred to a secure excel document. The excel document will be password protected. Paper forms will be placed in a secure cabinet in a locked office. Only members of the research team will have access to the electronic and paper forms.

5. Risk Assessment The risks associated with bicaval cannulation are minimal. There is potential for increased risk of bleeding because of the need for two incisions instead of one. Since we're cannulating the SVC and IVC indirectly through atrial incisions these potential bleeding sites can be easily seen and controlled intra-operatively.

There is a possibility of increased incidence of atrial fibrillation post-operatively in the intervention group. Although uncommon, some surgeons routinely perform bicaval cannulation for CABG.

Participants may benefit from the intervention if it leads to decreased rate of POAF. Thus avoiding the potential sequelae of AF and the side effects of treatment.

6. PUBLICATION We plan to use the data obtained in this study for publication in a peer-review journal. We may present the findings of the study in scientific conferences. No identifiable information will be published.

Appendix A: Consent form

Study Title: Effect of venous cannulation technique on the incidence of post-operative atrial fibrillation in patients undergoing elective coronary artery bypass grafting. A pilot randomized controlled trial.

Principle investigators: Jean-Francois Morin MD, Husain Esmaeil MD , Alex Alojko Study Site: Jewish General Hospital Address: 3755 Chemin de la Côte-Sainte-Catherine, Montréal, QC H3T 1E2 Telephone: (514) 340-8222

Introduction You are being asked to participate in a research study. Before agreeing to participate, it is important that you read the following explanation of this study.

The decision to participate in this study is up to you. Your participation is completely voluntary. Your decision will not affect your relationship with your regular doctor or your current or future medical care.

Please read this form carefully. Feel free to discuss the study with your family, friends, and healthcare provider before you make your decision whether to participate. Ask about anything you don't understand or would like explained better. Take time to decide whether or not you want to take part in this study and ask the study doctor or study staff as many questions about the study as you would like.

Background and purpose You are being asked to take part in this study because you have been diagnosed with coronary artery disease and will undergo coronary artery bypass grafting.

Atrial fibrillation is a type of heart arrhythmia that occurs in about 30% of patients undergoing coronary artery bypass grafting. This rhythm problem could cause a clot to form in the heart; this clot can travel to brain and cause a stroke. Atrial fibrillation is a treatable condition. The treatment method depends on the clinical situation. It is usually treated with medications that either controls the speed or the rhythm of the heart. If the arrhythmia causes severe symptoms such as chest pain, dizziness or hypotension (low blood pressure) it is sometimes treated with an electrical current (called electrical cardioversion) to restore the heart to its normal rhythm.

During heart surgery, the heart will be stopped in order to perform the coronary artery bypass surgery. The heart will be connected to a heart-lung machine (also called cardiopulmonary bypass machine). This machine takes over the job of the heart and lungs. A plastic tube will be connected to right upper chamber of the heart (called the right atrium) to the machine (this tube is called the venous cannula); the tube carries blood from the heart into an oxygenator where it will be oxygenated. The oxygenated blood is pumped into the body through a tube connected to the aorta (the body's main blood vessel).

Another method of the venous cannulation is by connecting two tubes to the superior vena cava and inferior vena cava (the two major veins carrying blood returning from the body to the right atrium of the heart). This is the same method used for mitral and tricuspid valve operations.

The purpose of this study is to look into the effect of different venous cannulation methods on the occurrence of atrial fibrillation (a type of arrhythmia) post coronary artery bypass grafting. This study has 2 groups. You will be randomly assigned to one of the two groups. The first group will have the venous cannula connected to the right atrium (which is the standard method). The second group will have the venous cannula connected to the superior and inferior vena cava and a tie is secured around the cannula so that no blood passes into the right atrium instead, the blood goes to the heart-lung machine.

Potential Risks

There are potential risks to you by taking part in this study. The rate of occurrence of atrial fibrillation (heart arrhythmia) could be higher in the treatment group you are assigned to. The bleeding risk is theoretically higher since we are making an incision in 2 areas to insert the cannulas instead of a single incision in the standard method. If bleeding occurs, you might need a blood transfusion or in uncommonly, you might need to be re-operated on to control the bleeding. In addition, there are some risks inherent to the coronary artery bypass grafting surgery, which include bleeding, heart attack, heart rhythm problems, heart failure (which is inadequate pumping of blood by the heart). Depending on the cause of the heart attack, It can be managed with medications, going back to surgery or by coronary angioplasty and placing a stent. Heart failure is treated with medications.

Other potential risks of coronary artery bypass grafting include liver problems (elevated liver enzymes due to inadequate blood supply during the operation), kidney injury (due to inadequate blood supply during the operation). Liver and kidney complications are usually managed with monitoring of their functions.

Other risks inherent to the surgery include lung problems such as lung infection, fluid collecting in the lungs or inability to disconnect the ventilator machine after the operation due to inability of the lungs to oxygenate the blood on their own and other uncommon risks such as stroke and death.

Potential Benefits

You may benefit as a result of your participation in this study. The rate of atrial fibrillation could be lower in the treatment group you are assigned to. However, there is no assurance that you will benefit from your participation in this study. Results from this study may benefit other patients in the future.

Alternative Treatments

This clinical study is for research purposes only. You do not have to participate in the study to receive treatment for coronary artery disease. The other option is a standard venous cannulation method in which the right atrium is cannulated.

Voluntary Participation/Withdrawal Your decision to participate in this clinical research study is voluntary. You may choose not to participate or you may withdraw from the study for any reason at any time without penalty. You should tell the study doctor or study team if you decide to leave the study.

The study doctor can stop the study or your participation in the study at any time without your consent if it appears to be medically harmful to you, if the study is cancelled, or for administrative reasons.

Confidentiality As part of this research, we will collect personal information from you (this means information that can identify you). In order to protect your privacy, all information collected will remain confidential to the extent permitted by law. Your identifiable health information is protected by a law. If the results of this study are published or presented at meetings, you will not be identified.

For monitoring, control, protection and security purposes, your research study file could be checked by persons authorized by the Research Ethics Committee of the CIUSSS du Centre-Ouest-de-l'Île de Montréal. These persons are bound by a confidentiality agreement.

For all questions concerning your rights during your participation in this study, or if you have any complaints or comments regarding your experience in taking part in this research study, you can contact the Local Commissioner of Complaints and Quality of Service of the CIUSSS Centre-Ouest-de-l'Île-de-Montréal or the ombudsman of the institution at (514) 340-8222, ex. 24222.

STATEMENT OF CONSENT

Study title: Effect of venous cannulation technique on the incidence of post-operative atrial fibrillation in patients undergoing elective coronary artery bypass grafting. A pilot randomized controlled trial.

PARTICIPANT STATEMENT

I understand the information that was explained to me as contained in this consent form. All my questions were answered to my satisfaction. I will receive a copy of this signed consent form. My participation is voluntary and I can withdraw from the research study at any time without any consequences and without having to give a reason. Withdrawing from this research study, at any time, will not affect my medical care now, or later, in any way. By signing this consent form, I do not give up any of my legal rights.

I agree to participate in this research study.

Name of Participant

Signature Date

RESEARCHER STATEMENT

I, as the person obtaining consent, certify that I have explained to the participant or his/her legal representative (where applicable) the research study information contained in this consent form and have answered all questions. I have clearly explained to the participant that s/he is free to withdraw at any time without providing a reason, and without any consequences. I commit, together with the members of the research team to respect all conditions described in this consent form and to give a signed copy of the consent form to the participant.

Name and signature of the researcher or person delegated to obtained consent

Date

Translator/Witness (if applicable)

Name and signature of translator/witness Date

ELIGIBILITY:
Inclusion Criteria:

Patients admitted for coronary artery bypass grafting under the care of the principal investigator at the Jewish General Hospital during the study period will be included if they meet all the following criteria:

1. Age >18 years
2. Sinus rhythm with HR >50bpm
3. Scheduled to undergo isolated elective on-pump CABG
4. Hemodynamically stable.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Second or third degree heart block
2. LVEF <35%
3. left atrial volume index ≥42 ml/m2
4. right atrial volume index > 47 ml/m2
5. any degree of tricuspid regurgitation
6. any degree of right ventricular dysfunction
7. emergency or minimally invasive operation
8. concurrent valve operation
9. history of atrial fibrillation
10. previous cardiac surgery
11. previous catheter ablation for atrial fibrillation
12. pre-operative use of class I or III anti-arrhythmics.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation | During hospital admission and clinic visit at 30 days from hospital discharge date.
  Number of participants who develop atrial fibrillation that requires treatment. Atrial fibrillation will be defined as any episode in any participant lasting >5 minutes in duration or any episode leading to hemodynamic compromise (SBP<90 mmHg) or causing symptoms (angina or dyspnea).

SECONDARY OUTCOMES:
Tricuspid regurgitation | on transthoracic echocardiogram performed on day 2-5 post-operatively
  Number of participants who develop any degree of tricuspid regurgitation
Right ventricular dysfunction | on transthoracic echocardiogram performed on day 2-5 post-operatively
  Number of participants who develop any degree of right ventricular dysfunction
Increase in Left atrial index | on transthoracic echocardiogram performed on day 2-5 post-operatively
  Number of participants who have an increase in left atrial volume index post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Morin, MD,FRCSC, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maesen B, Nijs J, Maessen J, Allessie M, Schotten U. Post-operative atrial fibrillation: a maze of mechanisms. Europace. 2012 Feb;14(2):159-74. doi: 10.1093/europace/eur208. Epub 2011 Aug 6. PMID 21821851
- [Background] Attaran S, Shaw M, Bond L, Pullan MD, Fabri BM. Atrial fibrillation postcardiac surgery: a common but a morbid complication. Interact Cardiovasc Thorac Surg. 2011 May;12(5):772-7. doi: 10.1510/icvts.2010.243782. Epub 2011 Feb 28. PMID 21357310
- [Background] Mariscalco G, Klersy C, Zanobini M, Banach M, Ferrarese S, Borsani P, Cantore C, Biglioli P, Sala A. Atrial fibrillation after isolated coronary surgery affects late survival. Circulation. 2008 Oct 14;118(16):1612-8. doi: 10.1161/CIRCULATIONAHA.108.777789. Epub 2008 Sep 29. PMID 18824644
- [Background] Filardo G, Hamilton C, Hebeler RF Jr, Hamman B, Grayburn P. New-onset postoperative atrial fibrillation after isolated coronary artery bypass graft surgery and long-term survival. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):164-9. doi: 10.1161/CIRCOUTCOMES.108.816843. Epub 2009 Apr 24. PMID 20031833
- [Background] Mathew JP, Fontes ML, Tudor IC, Ramsay J, Duke P, Mazer CD, Barash PG, Hsu PH, Mangano DT; Investigators of the Ischemia Research and Education Foundation; Multicenter Study of Perioperative Ischemia Research Group. A multicenter risk index for atrial fibrillation after cardiac surgery. JAMA. 2004 Apr 14;291(14):1720-9. doi: 10.1001/jama.291.14.1720. PMID 15082699
- [Background] Perrier S, Meyer N, Hoang Minh T, Announe T, Bentz J, Billaud P, Mommerot A, Mazzucotelli JP, Kindo M. Predictors of Atrial Fibrillation After Coronary Artery Bypass Grafting: A Bayesian Analysis. Ann Thorac Surg. 2017 Jan;103(1):92-97. doi: 10.1016/j.athoracsur.2016.05.115. Epub 2016 Aug 28. PMID 27577036
- [Background] Rousou JA, Meeran MK, Engelman RM, Breyer RH, Lemeshow S. Does the type of venous drainage or cardioplegia affect postoperative conduction and atrial arrhythmias? Circulation. 1985 Sep;72(3 Pt 2):II259-63. PMID 3875436
- [Background] Maisel WH, Rawn JD, Stevenson WG. Atrial fibrillation after cardiac surgery. Ann Intern Med. 2001 Dec 18;135(12):1061-73. doi: 10.7326/0003-4819-135-12-200112180-00010. PMID 11747385
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Schotten U, Verheule S, Kirchhof P, Goette A. Pathophysiological mechanisms of atrial fibrillation: a translational appraisal. Physiol Rev. 2011 Jan;91(1):265-325. doi: 10.1152/physrev.00031.2009. PMID 21248168
- [Background] Crystal E, Garfinkle MS, Connolly SS, Ginger TT, Sleik K, Yusuf SS. Interventions for preventing post-operative atrial fibrillation in patients undergoing heart surgery. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD003611. doi: 10.1002/14651858.CD003611.pub2. PMID 15495059
- [Background] Boos CJ, Anderson RA, Lip GY. Is atrial fibrillation an inflammatory disorder? Eur Heart J. 2006 Jan;27(2):136-49. doi: 10.1093/eurheartj/ehi645. Epub 2005 Nov 8. PMID 16278230
- [Background] Mathew JP, Parks R, Savino JS, Friedman AS, Koch C, Mangano DT, Browner WS. Atrial fibrillation following coronary artery bypass graft surgery: predictors, outcomes, and resource utilization. MultiCenter Study of Perioperative Ischemia Research Group. JAMA. 1996 Jul 24-31;276(4):300-6. PMID 8656542
- [Background] Amar D, Shi W, Hogue CW Jr, Zhang H, Passman RS, Thomas B, Bach PB, Damiano R, Thaler HT. Clinical prediction rule for atrial fibrillation after coronary artery bypass grafting. J Am Coll Cardiol. 2004 Sep 15;44(6):1248-53. doi: 10.1016/j.jacc.2004.05.078. PMID 15364327
- [Background] Chua SK, Shyu KG, Lu MJ, Lien LM, Lin CH, Chao HH, Lo HM. Clinical utility of CHADS2 and CHA2DS2-VASc scoring systems for predicting postoperative atrial fibrillation after cardiac surgery. J Thorac Cardiovasc Surg. 2013 Oct;146(4):919-926.e1. doi: 10.1016/j.jtcvs.2013.03.040. Epub 2013 Apr 26. PMID 23628495
- [Background] Khan AM, Lubitz SA, Sullivan LM, Sun JX, Levy D, Vasan RS, Magnani JW, Ellinor PT, Benjamin EJ, Wang TJ. Low serum magnesium and the development of atrial fibrillation in the community: the Framingham Heart Study. Circulation. 2013 Jan 1;127(1):33-8. doi: 10.1161/CIRCULATIONAHA.111.082511. Epub 2012 Nov 21. PMID 23172839
- [Background] Zaman AG, Archbold RA, Helft G, Paul EA, Curzen NP, Mills PG. Atrial fibrillation after coronary artery bypass surgery: a model for preoperative risk stratification. Circulation. 2000 Mar 28;101(12):1403-8. doi: 10.1161/01.cir.101.12.1403. PMID 10736284
- [Background] Booth JV, Phillips-Bute B, McCants CB, Podgoreanu MV, Smith PK, Mathew JP, Newman MF. Low serum magnesium level predicts major adverse cardiac events after coronary artery bypass graft surgery. Am Heart J. 2003 Jun;145(6):1108-13. doi: 10.1016/S0002-8703(03)00077-2. PMID 12796771
- [Background] Fairley JL, Zhang L, Glassford NJ, Bellomo R. Magnesium status and magnesium therapy in cardiac surgery: A systematic review and meta-analysis focusing on arrhythmia prevention. J Crit Care. 2017 Dec;42:69-77. doi: 10.1016/j.jcrc.2017.05.038. Epub 2017 Jun 21. PMID 28688240
- [Background] Lancaster TS, Schill MR, Greenberg JW, Moon MR, Schuessler RB, Damiano RJ Jr, Melby SJ. Potassium and Magnesium Supplementation Do Not Protect Against Atrial Fibrillation After Cardiac Operation: A Time-Matched Analysis. Ann Thorac Surg. 2016 Oct;102(4):1181-8. doi: 10.1016/j.athoracsur.2016.06.066. Epub 2016 Sep 2. PMID 27596917
- [Background] Cook RC, Yamashita MH, Kearns M, Ramanathan K, Gin K, Humphries KH. Prophylactic magnesium does not prevent atrial fibrillation after cardiac surgery: a meta-analysis. Ann Thorac Surg. 2013 Feb;95(2):533-41. doi: 10.1016/j.athoracsur.2012.09.008. Epub 2012 Nov 7. PMID 23141526
- [Background] Kalus JS, Caron MF, White CM, Mather JF, Gallagher R, Boden WE, Kluger J. Impact of fluid balance on incidence of atrial fibrillation after cardiothoracic surgery. Am J Cardiol. 2004 Dec 1;94(11):1423-5. doi: 10.1016/j.amjcard.2004.08.017. PMID 15566917
- [Background] Matsuura K, Ogino H, Matsuda H, Minatoya K, Sasaki H, Yagihara T, Kitamura S. Impact of volume status on the incidence of atrial fibrillation following aortic arch repair. Heart Vessels. 2007 Jan;22(1):21-4. doi: 10.1007/s00380-006-0928-y. Epub 2007 Jan 26. PMID 17285441
- [Background] Panesar SS, Athanasiou T, Nair S, Rao C, Jones C, Nicolaou M, Darzi A. Early outcomes in the elderly: a meta-analysis of 4921 patients undergoing coronary artery bypass grafting--comparison between off-pump and on-pump techniques. Heart. 2006 Dec;92(12):1808-16. doi: 10.1136/hrt.2006.088450. Epub 2006 Jun 14. PMID 16775087
- [Background] Tchervenkov CI, Wynands JE, Symes JF, Malcolm ID, Dobell AR, Morin JE. Persistent atrial activity during cardioplegic arrest: a possible factor in the etiology of postoperative supraventricular tachyarrhythmias. Ann Thorac Surg. 1983 Oct;36(4):437-43. doi: 10.1016/s0003-4975(10)60484-5. PMID 6605126
- [Background] Rosenfeldt FL, Watson DA. II. Interference with local myocardial cooling by heat gain during aortic cross-clamping. Ann Thorac Surg. 1979 Jan;27(1):13-6. doi: 10.1016/s0003-4975(10)62964-5. PMID 453953
- [Background] Bennett EV Jr, Fewel JG, Grover FL, Trinkle JK. Myocardial preservation: effect of venous drainage. Ann Thorac Surg. 1983 Aug;36(2):132-42. doi: 10.1016/s0003-4975(10)60446-8. PMID 6882072